CLINICAL TRIAL: NCT05291273
Title: Influence of Anthropometric Data, Shoulder Complex Muscle Strength, and Abdominal-lumbar Endurance in Closed Kinetic Chain Upper Extremity Stability Test
Acronym: EPOLTEST 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC22.0005
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Pain
Keywords: CKCUEST; Physical activity; Rehabilitation
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a monocentric interventional prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All subjects will perform the same tests.
  Interventions: Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Prone Bridge Test; Diagnostic Test: Measurement of the muscle strength of the shoulder complex

INTERVENTIONS:
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — Each patient receive the same intervention, the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST). The CKCUEST is a functional test which assess shoulder's stability. Patient is in push-up position, with 91 cm between his hands. His body is straight and his foots are squeeze. patient has to touch his hand with his other one and returns in the initial position. Then, patient repeats this movement with his other hand, etc, during 15 secondes. The CKCUEST score is the movement's number performed.
Diagnostic Test: Prone Bridge Test — The prone bridge test also known as the "plank" or "hover" measures the muscular endurance of the abdominal muscles. Subjects will start in the "down" push up position with their feet together and their hands shoulder width apart. When the test starts the subject will push up to the prone bridge position so they are resting on their hands and toes making sure they maintain a straight line from the shoulders through the hips to the knees. The outcome measure will be the time where the subject stay in this position.
Diagnostic Test: Measurement of the muscle strength of the shoulder complex — Maximum isometric force of the external and internal rotators and abductors/adductors measured by a dynamometer.

SUMMARY:
A previous study of the Closed Kinetic Chain Upper Extremity Stability Test (EPOLTEST) in a population aged 18 to 25 years isolated 3 main factors influencing the CKCUEST score: upper extremity span, weight, and sex of the individual. A predictive equation for the CKCUEST score was thus established and to date has a capacity to determine the real score of approximately 51%.

The results of this first study show that a certain number of variables have not been studied.

The purpose of this study, EPOLTEST 2, is to take into account the variables already studied on a larger population (18-50 years old) and to add an assessment of shoulder muscle strength and abdominolumbar endurance.

ELIGIBILITY:
Inclusion Criteria:

* Aged to 18 to 50 years
* Capacity to consent
* Who has signed the consent

Exclusion Criteria:

* Fracture history or upper limb luxation < 1 year
* Pain or discomfort that prevents the test from being performed
* History of abdominal surgery or hernia < 1 year
* Pregnant or nursing
* Refuse to participate
* Guardianship or protection of vulnerable adult

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 247 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) score | Day 1
  Closed Kinetic Chain Upper Extremity Stability Test/ The CKCUEST is a functional test which assess shoulder's stability. Patient is in push-up position, with 91 cm between his hands. His body is straight and his foots are squeeze. Patient has to touch his hand with his other one and returns in the initial position. Then, patient repeats this movement with his other hand, etc, during 15 secondes. The CKCUEST score is the movement's number performed. Three tests are performed. The outcome measure will be the mean of the score of the three tests realisation.
Anthropometric data | Day 1
  Measurement of the subject's weight in kilograms
Anthropometric data | Day 1
  Measurement of the subject's height in centimeters
Anthropometric data | Day 1
  Measurement of the subject's BMI in kg/m^2
Anthropometric data | Day 1
  Measurement of the subject's upper extremity length in centimeters
Anthropometric data | Day 1
  Measurement of the subject's upper extremity span in centimeters
Anthropometric data | Day 1
  Measurement of the subject's distance between acromion and radial styloid of the right upper limb in centimeters
Anthropometric data | Day 1
  Measurement of the subject's distance between olecranon and radial styloid of the right upper limb in centimeters
Muscular strength of the shoulder complex | Day 1
  Maximum isometric force of the external and internal rotators and abductors/adductors measured by a dynamometer in Newton.
Abdominal-lumbar stability | Day 1
  The prone bridge test also known as the "plank" or "hover" measures the muscular endurance of the abdominal muscles. Subjects will start in the "down" push up position with their feet together and their hands shoulder width apart. When the test starts the subject will push up to the prone bridge position so they are resting on their hands and toes making sure they maintain a straight line from the shoulders through the hips to the knees. The outcome measure will be the time where the subject stay in this position.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.